CLINICAL TRIAL: NCT06082284
Title: A Cross-sectional Study on the Positive Rate of Monoclonal Immunoglobulin (M Protein) in the Serum of Patients Seeking Medical Treatment in Tertiary Hospitals Based on a Highly Sensitive Serum M Protein Detection Method.
Brief Title: A Cross-sectional Study on the Positive Rate of M Protein Based on a Highly Sensitive Serum M Protein Detection Method.
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhujiangzny
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma; M Protein
Keywords: M protein
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who come to the hospital for treatment: Patients attending the outpatient/emergency/inpatient department of Zhujiang Hospital over 18 years old.

SUMMARY:
By using a highly sensitive serum M protein detection method based on the MALDI-TOF MS platform, serum monoclonal immunoglobul (M protein) in detection was performed on the visiting patients to explore the positive rate of serum M protein and its distribution in different departments. And exploring the correlation analysis between the relative concentration of serum M protein based on the above highly sensitive methods and clinical indicators.

DETAILED DESCRIPTION:
Monoclonal gammopathy (MG) is an asymptomatic pre-cancerous clonal proliferation of plasma cells. The onset of this disease is concealed, usually discovered by chance by patients who undergo protein electrophoresis to detect monoclonal gamma globulin (M protein) due to various clinical symptoms and disease evaluations. Due to the insidious onset of monoclonal immunoglobulin, involving multiple organs, and the non-specific clinical symptoms, it is more prone to misdiagnosis. This study hypothesized that among patients who first came to the hospital for treatment, some patients had elevated serum monoclonal immunoglobulin levels but were not initially diagnosed with hematology department, but instead sought medical attention from other departments due to other symptoms. In this study，by using a highly sensitive serum M protein detection method based on the MALDI-TOF MS platform, serum monoclonal immunoglobul (M protein) in detection was performed on the visiting patients to explore the positive rate of serum M protein and its distribution in different departments，and to explore the correlation analysis between the relative concentration of serum M protein based on the above highly sensitive methods and clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the outpatient/emergency/inpatient department of Zhujiang Hospital;
* Age: over 18 years old;
* There are sufficient remaining serum samples and extensive informed consent has been signed.

Exclusion Criteria:

* Early diagnosis of hematological diseases such as plasma cell or other B lymphocyte proliferative diseases；
* Improper storage or repeated freeze-thaw of remaining serum samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old attending the outpatient/emergency/inpatient departments of Zhujiang Hospital, including departments such as hematology, general surgery, dermatology, and others.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive rate of M protein | one year
  Positive rate of serum M protein in patients seeking medical treatment at the hospital
The distribution of positive rate of M protein in different departments | one year
  The positive rate of serum M protein in the patients visiting the hospital and its distribution in different departments.

SECONDARY OUTCOMES:
Correlation analysis | one year
  Correlation analysis between the relative concentration of serum M protein and clinical indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No